CLINICAL TRIAL: NCT01544218
Title: Validating NIAAA's Brief Screening Guide in Youth With Chronic Medical Conditions
Brief Title: Validating NIAAA Screen Guide in YCMC
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sharon Levy, Assistant Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: SL_NIAAARFA_0212
Record Dates: First submitted 2012-02-15; First posted 2012-03-05 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Alcohol Related Disorders
Keywords: Alcohol related disorders
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- YCMC: Youth ages 9-18 with one of four chronic medical conditions - asthma, diabetes, rheumatic or gastroenterologic conditions

SUMMARY:
Alcohol use is a serious health threat to the 26% youth in the US with chronic medical conditions. While alcohol use can significantly impact an underlying illness and its safe/effective management, medical specialists rarely screen their adolescent patients for alcohol use. The investigators will validate a new, brief alcohol- screening tool with 9-18 year old youth with chronic medical conditions. Comprehensive assessment information will be collected and analyzed to describe relationships between youth alcohol use, other substance use, and chronic disease outcomes and findings integrated into the validated screen as actionable clinician guidance and health advice.

ELIGIBILITY:
Inclusion Criteria:

* 9-18 years of age
* duration of chronic illness of at least one year
* ability to speak/read English and use a computer keyboard and/or complete an interviewer-assisted questionnaire

Exclusion Criteria:

* medically or emotionally unstable
* unable to assent/consent

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 9-18 year old youth with one of four chronic conditions - asthma, diabetes, rheumatic or gastroenterologic conditions
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07-20 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
eGuide diagnosis of alcohol use disorder | Baseline
  We will evaluate the sensitivity and specificity of the eGuide to correctly identify the group of YCMC who have problem use/abuse or dependence, using the CIDI-SAM as the criterion standard.

SECONDARY OUTCOMES:
Correlation of HgbA1c level with level of alcohol use | Baseline
Correlation between score on the Asthma Control Test (ACT)and level of alcohol use | Baseline
Correlation of score on The Childhood Health Assessment Questionnaire (CHAQ) with level of alcohol use | baseline
Correlation between The Pediatric Ulcerative Colitis Activity Index (PUCAI)score and level of alcohol use | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, MPH, Principal Investigator — Boston Children's Hospital; Elissa Weitzman, ScD, MSc, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States